CLINICAL TRIAL: NCT03046953
Title: A Phase 2a Trial of Avelumab, an Anti-PDL1 Antibody, in Relapsed and Refractory Peripheral T-cell Lymphoma
Brief Title: Avelumab in Relapsed and Refractory Peripheral T-cell Lymphoma
Acronym: AVAIL-T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Bloodwise (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_16-123
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: T-Cell Lymphoma Relapsed; T-Cell Lymphoma Refractory
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: Single Arm trial with bayesian design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): Avelumab 10mg/kg by IV infusion once every 2 weeks. A maximum of 8 cycles, each cycle is 28 days.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — anti-PDL1 antibody
  Other Names: MSB0010718C

SUMMARY:
The AVAIL-T trial is a trial to find out how effective avelumab is at treating patients with primary T-cell lymphoma that is refractory to or has relapsed following initial treatment.

DETAILED DESCRIPTION:
The AVAIL-T trial is designed to find out how effective avelumab is at treating patients with primary T-cell lymphoma that is refractory to or has relapsed following initial treatment. Up to 36 people will be taking part in the AVAIL-T trial at hospitals across the United Kingdom. All patients on the trial will be recruited over 2 years and receive up to 8 cycles of avelumab treatment. Avelumab is an anti-PDL1 (programmed cell death receptor ligand 1) antibody that will be given as an infusion once every 2 weeks in cycles lasting 28 days. The trial will be looking at the response to avelumab, by measuring the change in the tumour size using CT scans, and seeing how long that response is maintained. The trial will also look at toxicity, overall survival, and progression free survival.

In addition we will analyse blood samples and samples of the cancer to understand better how the cancer behaves. This may guide the investigators in developing better treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 16 years
* Life expectancy > 12 weeks
* ECOG (eastern oncology cooperative group) performance status ≤ 2
* Relapsed or refractory* peripheral T-cell lymphoma including the following histologies: peripheral T-cell lymphoma not otherwise specified (PTCL NOS) , angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL), enteropathy associated T-cell lymphoma (EATL), extranodal NK (natural killer)/T- cell lymphoma (ENKL), transformed mycosis fungoides (LCT MF), hepatosplenic T-cell lymphoma (HSTCL) * For all relapsed patients, relapse must be confirmed by tissue biopsy (or bone marrow trephine if no other tissue available). For refractory patients, a biopsy must have been obtained within the last 3 months
* Failed at least 1 prior therapy (but no upper limit of prior regimens)
* Adequate haematological function defined by at registration:

  * absolute neutrophil count (ANC) ≥ 1.0 × 109/L, (unsupported)
  * platelet count ≥ 75 × 109/L, (unsupported)
  * haemoglobin ≥ 9 g/dL (may have been transfused)
* Adequate hepatic function defined by:

  * total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range
  * AST (aspartate aminotransferase) or ALT (alanine aminotransferase) levels ≤ 2.5 × ULN for all patients, or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver)
* Adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
* CT measurable disease with at least 1 lesion having short axis > 1.5cm or splenomegaly > 14cm in cranio-caudal length attributable to relapsed/non responding lymphoma
* Negative serum pregnancy test at screening for women of childbearing potential.
* Highly effective contraception for both male and female patients if the risk of conception exists. (Note: women of childbearing potential and men able to father a child must agree to use 2 highly effective contraception, defined as methods with a failure rate of less than 1 % per year. Highly effective contraception is required from consent, throughout and for at least 60 days after avelumab treatment.
* Ability to give informed consent

Exclusion Criteria:

Patients are not eligible for the trial if they fulfill any of the following exclusion criteria:

* All patients with active central nervous system (CNS) involvement of lymphoma
* Prior organ transplantation, including allogeneic stem cell transplantation
* Significant acute or chronic infections including, among others:

  * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS),
  * Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* Current use of immunosuppressive medication, EXCEPT for the following:

  * intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); Systemic corticosteroids at a maximum dose of ≤ 1 mg/kg of prednisone or equivalent during screening (to be stopped by day 1 of trial treatment); Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy Grade ≤ 2 or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable are acceptable
* Pregnancy or lactation
* Known alcohol or drug abuse
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to registration), myocardial infarction (< 6 months prior to registration), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
* Active infection requiring systemic therapy
* Major surgery within 4 weeks of trial entry
* Patients and partners of childbearing potential not willing to use two methods of effective contraception during and for 60 days after therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Wagner, MD, Principal Investigator — Univeristy of Leicester
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited from November 14, 2017 to November 18, 2019 at 14 UK (United Kingdom) hospitals by clinician referral. The first patient was recruited on December 8, 2017, and the final patient recruited on November 18, 2019.
Pre-assignment Details: Of 35 enrolled patients, only 32 started treatment. Of the 3 patients who did not start treatment, one died, one relapsed and one was found to be ineligible post registration.
Groups:
- Avelumab: Patients received Avelumab 10mg/kg by IV infusion once every 2 weeks. A maximum of 8 cycles, each cycle is 28 days.
  Avelumab: anti-PDL1 antibody
Period: Overall Study
Arm/Group | Avelumab
Started | 32 (Of the 35 patients registered on the trial, only 32 actually started treatment.)
Completed Cycle 3 (Patients had to reach the CT scan assessment for cycle 3 to be evaluable for the trial) | 16 (16 patients completed cycle 3 with disease assessments done and so were evaluable)
Completed Cycle 6 | 10 (10 patients completed cycle 6, 9 disease assessments done, one disease assessment not done)
Completed Cycle 8 | 6 (6 patients completed cycle 8, 4 disease assessments done, 2 disease assessments not done)
Completed | 6
Not Completed | 26
Not completed — Relapse/progressive disease | 21
Not completed — Death | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Intention to treat population was 35
Arm/Group | Avelumab
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Histology [Count of Participants; unit: Participants]
  Peripheral T-cell lymphoma not otherwise specified | 17
  Angioimmunoblastic T-cell lymphoma | 11
  Extranodal NK/T-cell lymphoma | 4
  Anaplastic large cell lymphoma | 1
  Transformed mycosis fungoides | 1
  Missing data | 1
Prior therapies [Median (Inter-Quartile Range); unit: years] | 3.0 [2.0 to 3.0]
ECOG performance [Count of Participants; unit: Participants] — GRADE ECOG PERFORMANCE STATUS
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 17
    1 | 13
    2 | 4
    Missing Data | 1
Weight [Mean (Standard Deviation); unit: kg] — Includes all patients eligible at registration Population: 1 patient ineligible post registration
  kg
    number analyzed (Participants) | 34
    (all) | 81.7 (17.3)
Height [Mean (Standard Deviation); unit: metres] — Includes all patients eligible at registration Population: 1 patient was ineligible post registration
  metres
    number analyzed (Participants) | 34
    (all) | 1.7 (0.1)
BMI [Mean (Standard Deviation); unit: kg/m2] — Includes all patients eligible at registration Population: 1 patient was ineligible post registration
  kg/m2
    number analyzed (Participants) | 34
    (all) | 27.0 (5.1)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Includes all patients eligible at registration Population: 1 patient was ineligible post registration
  mmHg
    number analyzed (Participants) | 34
    (all) | 127.0 (19.7)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Includes all patients eligible at registration Population: 1 patient was ineligible post registration
  mmHg
    number analyzed (Participants) | 34
    (all) | 74.2 (9.8)
Pulse [Mean (Standard Deviation); unit: bpm] — Includes all patients eligible at registration Population: 1 patient was ineligible post registration
  bpm
    number analyzed (Participants) | 34
    (all) | 83.7 (21.7)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate During the First 8 Cycles of Treatment
Description: Best overall response rate (Completed response [CR] + partial remission [PR]) during the first 8 cycles of treatment will be assessed using contrast-enhanced CT scans of the neck, chest, abdomen and pelvis, using the Revised Response Criteria for Malignant Lymphoma. In this study CR = complete disappearance of all detectable clinical evidence of disease, so involved lymph nodes had regressed on CT scan to normal size. PR = al least a 50% decrease in size of the involved lymph nodes measured on CT scans.
Time Frame: 8 cycles (224 days)
Population: The per-protocol population was used ,defined as all patients recruited to the trial who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 32
Participants | 5

2. Secondary Outcome: Toxicity- Number of Patients
Description: Toxicity assessed using CTCAE v4.0 will be defined as the number of patients who experience one or more grade 3 or 4 adverse event or serious adverse event of any grade
Time Frame: During treatment of 8 cycles (224 days)
Population: The number of patients in the per-protocol population who experience one or more grade 3 or 4 adverse event or serious adverse event of any grade
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 32
Participants | 21

3. Secondary Outcome: Toxicity- Proportion of Patients
Description: Toxicity assessed using CTCAE v4.0 will be defined as the proportion of patients who experience one or more grade 3 or 4 adverse event or serious adverse event of any grade
Time Frame: During treatment of 8 cycles (224 days)
Population: The proportion of patients in the per-protocol population who experience one or more grade 3 or 4 adverse event or serious adverse event of any grade
Measure: Number; unit: proportion of patients
Arm/Group | Avelumab
Number analyzed (Participants) | 32
proportion of patients | 0.656

4. Secondary Outcome: Maximum Percentage Change in Sum of Product of Diameters
Description: Maximum percentage change in the sum of the product of diameters (SPD) of target tumour masses assessed by contrast-enhanced CT scans of the neck, chest, abdomen and pelvis, using the Revised Response Criteria for Malignant Lymphoma.
Time Frame: During trial treatment of 8 cycles (224 days), comparing baseline with cycles 3, 6 and 8
Population: 13 of the 32 patients who started treatment had available CT scans containing the target lesions at cycles 3, 6 or 8 for comparison with baseline, and these patients were included in this analysis
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Avelumab
Number analyzed (Participants) | 13
percentage change | -4.3 [-56.6 to 28.1]

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from first documented response (CR or PR) until relapse/progression, as determined by the Revised Response Criteria, or death. Patients who are relapse/progression free and alive at time of final analysis will be censored at date last seen.
Time Frame: 2 years
Population: Patients who responded
Measure: Median (Full Range); unit: months
Arm/Group | Avelumab
Number analyzed (Participants) | 5
months | 13.3 [6.8 to 23.2]

6. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from date of registration to the date of disease progression or date of death from any cause. Patients not reaching progression or death at the time of analysis will be censored at the last date they were known to be alive and progression free.
Time Frame: 2 years
Population: Per-protocol population defined as all patients recruited to the trial who started treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab
Number analyzed (Participants) | 32
months | 2.86 [1.77 to 4.37]

7. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from date of registration to the date of death from any cause. Patients discontinuing the study, lost to follow-up or still alive at the end of the study will be censored at the date of last follow-up.
Time Frame: Deaths were collected up to 2 years
Population: Per-protocol population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab
Number analyzed (Participants) | 32
months | 10.41 [6.60 to 12.25]

ADVERSE EVENTS:
Time Frame: Serious and other (not including serious) adverse events were recorded for all patients from the date they started trial treatment until 30 days after they received their last treatment, up to 9 months. Deaths were collected up to 2 years.
Description: Safety data for this trial was collected in accordance with CTCAE criteria version 4.0
Groups:
- Avelumab: Avelumab (an anti-PDL1 antibody) 10mg/kg by IV infusion once every 2 weeks. A maximum of 8 cycles, each cycle is 28 days.
Arm/Group | Avelumab
All-Cause Mortality (participants affected / at risk) | 24/32
Serious Adverse Events (participants affected / at risk) | 18/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Dacrocystitis (Eye disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Immune-mediated colitis (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 4 (6)
Infusion related reaction (General disorders) | 1 (1)
Edema-groin,scrotum (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Lung/skin infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Infection (blood culture positive) (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2)
Rhinitis infective (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Infections and infestations-Other,specify (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Mucositis Oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 5 (7)
Chills (General disorders) | 3 (3)
Edema Limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 8 (12)
Fever (General disorders) | 8 (11)
Flu Like Symptoms (General disorders) | 2 (2)
Infusion Related Reaction (General disorders) | 7 (7)
Localised Edema (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 4 (5)
Sepsis (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 2 (4)
Alkaline Phosphatase increased (Investigations) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 2 (2)
Platelet Count Decreased (Investigations) | 5 (11)
Weight Loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (8)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Lethargy (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
For one of the secondary outcomes- the maximum percentage change in the sum of the products of diameters, calculated from measurements of target tumour masses assessed by CT scans- no reliable conclusions could be drawn from this analysis due to missing data and a lack of consistent reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03046953/Prot_SAP_000.pdf